CLINICAL TRIAL: NCT02800785
Title: The Comparison of Outcomes of Antibiotic Drugs and Appendectomy (CODA) Trial
Acronym: CODA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, David Flum, Professor, Surgery, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001155
Record Dates: First submitted 2016-04-08; First posted 2016-06-15 (Estimated); Results first posted 2023-04-18 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Cefoxitin; Ertapenem; Moxifloxacin; Tigecycline; ticarcillin-clavulanic acid; Metronidazole; Cefazolin; Cefuroxime; Ceftriaxone; Cefotaxime; Ciprofloxacin; Levofloxacin; Appendectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antibiotics Therapy Arm (Active Comparator): Patients in the antibiotics (abx) arm will receive a total of 10 days of abx, with a minimum of 24 hours using an IV abx formulation (administered in q8, q12, or q24 hour regimens with or without concurrent oral abx) followed by oral abx for the remainder of the 10 days. Patients will be offered a treatment regimen of abx based on guidelines published jointly by the Surgical Infection Society and the Infectious Disease Society of America. Any of the IV abx options (Single antibiotic-Cefoxitin, Ertapenem, Moxifloxicin, Tigecycline, Ticarcillin-Clavulanic Acid or Dual antibiotics-Metronidazole plus one of the following-Cefazolin, Cefuroxime, Ceftriaxone, Cefotaxime, Ciprofloxacin, Levofloxacin) will be considered acceptable. After IV abx, a regimen of oral abx will be continued for a total treatment length of 10 days.
  Interventions: Drug: Cefoxitin, Ertapenem, Moxifloxacin, Tigecycline, Ticarcillin-Clavulanic Acid; Metronidazole plus Cefazolin, Cefuroxime, Ceftriaxone, Cefotaxime, Ciprofloxacin, or Levofloxacin
- Appendectomy Arm (Active Comparator): Patients in the appendectomy arm will have an appendectomy performed by an open or laparoscopic approach, depending on patient and surgeon preference. Prior to their operation, patients in this arm will receive one dose of antibiotics per currently accepted standards when appendicitis diagnosis is confirmed. Patients may also receive preoperative antibiotics per hospital standards for surgical infection prevention bundle.
  Interventions: Procedure: Appendectomy

INTERVENTIONS:
Drug: Cefoxitin, Ertapenem, Moxifloxacin, Tigecycline, Ticarcillin-Clavulanic Acid; Metronidazole plus Cefazolin, Cefuroxime, Ceftriaxone, Cefotaxime, Ciprofloxacin, or Levofloxacin — Patients will be offered a treatment regimen of antibiotics based on guidelines published jointly by the Surgical Infection Society and the Infectious Disease Society of America. After IV antibiotics are administered for a period of at least 24 hours, a regimen of oral antibiotics will be continued for a total treatment length of 10 days. Preferred oral antibiotic regimens include Moxifloxacin alone, and combinations such as Metronidazole or Clindamycin, for anaerobic bacteria coverage, plus Ciprofloxacin or Levofloxacin, or an oral Cephalosporin for aerobic Gram-negative bacteria coverage.
  Arms: Antibiotics Therapy Arm
Procedure: Appendectomy — Appendectomy will be performed by an open or laparoscopic approach, depending on patient and surgeon preference.
  Arms: Appendectomy Arm

SUMMARY:
For the past 130 years, appendectomy has been the standard treatment for appendicitis. Recent studies from Europe have challenged the notion that surgery is the best option, showing that antibiotics alone can treat appendicitis without a need for appendectomy in as many as 3 out of 4 patients and without safety issues for up to one year of follow up. Despite these results, it remains to be determined if the antibiotic strategy is as good as an appendectomy for the outcomes that most patients care about. The Patient-Centered Outcomes Research Institute (PCORI)-funded Comparison of Outcomes of Drugs and Appendectomy (CODA) trial will be the first American, and largest-ever randomized trial of the issue and its results should help surgeons and patients make more informed healthcare decisions.

DETAILED DESCRIPTION:
The Comparison of Outcomes of Antibiotic Drugs and Appendectomy (CODA) trial aims to test, if from a patient's perspective, the antibiotics strategy is "just as good as" surgery. The investigators believe that patients, clinicians, and the people who pay for healthcare (both patients and insurers) will find the antibiotics approach acceptable if 1) it results in high rates of treatment success, 2) does not increase complications, and 3) provides an equivalent or better patient experience. A large-scale non-inferiority trial is expected to result in a change in the management of one of the most common human illnesses. If non-inferiority is demonstrated (or superiority of the antibiotics approach identified), that finding will improve patient choice and should support a shift to the less invasive approach. If non-inferiority is not established, results may help to delineate the trade-offs between the two treatment approaches and inform decision-making.

The observation that patients with acute uncomplicated appendicitis (AUA) can be cured with antibiotics-alone has a scientific rationale. Traditionally, appendicitis was thought to result from a blockage of the appendix and that, if left untreated, inevitably led to a perforation. Contrary to this physiologic model, Carr demonstrated that obstruction of the appendix is an unlikely primary cause in the majority of patients and that most are caused by an enteric infection. A recent randomized trial found an increased rate of appendectomy with early use of computed tomography (CT) imaging and diagnostic laparoscopy, but case reports of appendicitis remission documented by serial CT all suggest that leaving the appendix in place does not inexorably lead to clinical compromise. A common concern of clinicians when considering treating AUA with antibiotics is that not removing the appendix may lead to perforation and complications from complicated appendicitis. Evidence suggests, however, that perforated appendicitis is a pre-hospital event and that non-perforated appendicitis is a "different" disease. This theory is supported by a general lack of relation between a delay in surgery of up to 24-36 hours and perforation rates. Most recently, Fusobacterium sp., a genus of enteric Gram-negative anaerobic bacteria, rather than an obstructive stone, was found to be correlated with the presence of appendicitis and the degree of inflammation. What remains to be determined is whether certain bacterial colonies or features of individual immune response are most associated with progression of appendicitis without appendectomy and whether successful outcomes for people undergoing antibiotics can be predicted based on the patient's characteristics.

An additional rationale for this study is to address limitations of prior trials. To avoid misclassification problems of other trials, all patients will undergo standard radiographic imaging including CT, ultrasound (US), or magnetic resonance imaging (MRI). Patients with an appendicolith will be included in the trial but considered a unique subgroup and will be evaluated as part of a pre-specified analysis (potentially excluding them from future recruitment if an early analysis demonstrates futility related to the primary antibiotic approach not being successful). To reflect usual and emerging techniques in treatment, the study includes both types of appendectomy (open and laparoscopic) and a broad range of antibiotic strategies including the option for an "all outpatient" treatment schedule with once daily dosing of longer-acting agents. Patients in the antibiotics arm will be given a minimum of 24 hours of intravenous (IV) antibiotics (using any appropriate dosing schedule and based on the patient's ability to tolerate oral medication), followed by oral antibiotics for a total of 10 days of antibiotic treatment). Discharge from the hospital or emergency department (ED) or a change in treatment arms will be guided by clinical targets and reasons for change in treatment arms will be assessed. Patients will be followed for up to two years to assess for longer-term complications, eventual appendectomy (performed anywhere), quality of life (QoL), gastrointestinal symptoms, and decisional regret. To quantify selection bias and to promote generalizability, all patients approached for the study and those who refuse randomization will be characterized at baseline. A parallel cohort of patients who refuse randomization (250 who initiate the antibiotics strategy and 250 who select the appendectomy strategy) will be surveyed for two years.

ELIGIBILITY:
Inclusion Criteria:

1. Adult ≥18 years;
2. Clinical diagnosis of acute uncomplicated appendicitis (AUA) established by clinical care team, supported by any of the following usual care radiological tests (computed tomography (CT), ultrasound (US), and/or magnetic resonance imaging (MRI)). AUA is defined by the usual signs, symptoms, and imaging finding of appendicitis without:

   1. Diffuse peritonitis on clinical exam (i.e., rigid abdomen / four quadrant peritonitis);
   2. Radiologic findings of :

   i. Free air; ii. Walled off fluid collection concerning for an abscess; iii. Significant amounts of intra-abdominal fluid throughout abdomen (i.e., more than trace fluid); or iv. Extent of inflammation or adjacent organ involvement on radiologic imaging such that appendectomy is relatively contraindicated.
3. Ability to provide written or electronic informed consent in English or Spanish.

Exclusion Criteria:

1. 1. Unable or unwilling to return or be contacted for clinical follow-up visits and/or research surveys;
2. Currently incarcerated in a detention facility or in police custody (patients wearing a monitoring device can be enrolled) at baseline/screening;
3. Evidence of severe sepsis or septic shock (e.g., new presumed sepsis-related organ dysfunction, elevated lactate, and/or fluid unresponsive hypotension);
4. Conditions with altered immune response or at risk for bacterial seeding;
5. Immunodeficiency (e.g., absolute neutrophil count <500/mm3, chronic immunosuppressive drugs, active chemotherapy or plans for chemotherapy in the following 30 days, or known acquired immune deficiency syndrome (AIDS) [cluster of differentiation 4 (CD4) count <200 or AIDS-defining illness within the last year] assessed by patient history);
6. Uncompensated liver failure;
7. Taking medication to treat active inflammatory bowel disease (e.g., Crohn's, ulcerative colitis);
8. Malignancy, not in remission (ongoing chemotherapy patients excluded);
9. Pregnant or expectation of becoming pregnant in the 30 days following baseline/screening;
10. Expected concurrent hemodialysis, peritoneal dialysis, or treatments using indwelling venous catheters;
11. Recent (within 90 days) placement of surgical implant (e.g., pacemaker, joint prosthesis, mechanical valve);
12. Indwelling Left Ventricular Assist Device (LVAD);
13. Patients with another infection (e.g., pneumonia, urinary tract infection) that requires treatment with another antibiotic at baseline/screening;
14. Concurrent illness that would otherwise mandate hospitalization outside of appendicitis and associated symptoms at baseline/screening;
15. Imaging findings of any of the following:

    1. Appendiceal soft-tissue mass;
    2. Imaging features of mucocele or tumor (e.g., appendix measuring ≥ 15mm in diameter and no other CT evidence of appendicitis);
    3. Concern for carcinomatosis on imaging; or
16. Severe allergy or reaction (e.g., immediate urticaria or anaphylaxis) to all of the proposed antibiotics;
17. Prior enrollment in the study or other investigational drug or vaccine while on study treatment;
18. Abdominal/pelvic surgery in the past month; or
19. More than seven hours have transpired since the patient received the first parenteral dose of antibiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1552 (Actual)
Dates: Start 2016-05; Primary Completion 2020-03-05 (Actual); Study Completion 2021-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Flum, MD, MPH, Principal Investigator — University of Washington; David A Talan, MD, Principal Investigator — University of California, Los Angeles
Locations (25):
- United States (25):
  - Olive View-UCLA Medical Center, Sylmar, California
  - Harbor-UCLA Medical Center, Torrance, California
  - University of Colorado Denver, Aurora, Colorado
  - Rush University Medical Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Maine Medical Center, Portland, Maine
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Michigan Medicine- University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - New York University - Bellevue Hospital, New York, New York
  - New York University - Tisch Hospital, New York, New York
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medicine, New York, New York
  - The Ohio State University Medical Center, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Lyndon B Johnson- Harris Health, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Providence Regional Medical Center Everett, Everett, Washington
  - Harborview Medical Center, Seattle, Washington
  - Virginia Mason University Village Medical Center, Seattle, Washington
  - Swedish Medical Center- First Hill, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Madigan Army Medical Center, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets, analytic datasets, and codebook will be shared back to study sponsor, PCORI.

REFERENCES:
- [Background] CODA Collaborative; Flum DR, Davidson GH, Monsell SE, Shapiro NI, Odom SR, Sanchez SE, Drake FT, Fischkoff K, Johnson J, Patton JH, Evans H, Cuschieri J, Sabbatini AK, Faine BA, Skeete DA, Liang MK, Sohn V, McGrane K, Kutcher ME, Chung B, Carter DW, Ayoung-Chee P, Chiang W, Rushing A, Steinberg S, Foster CS, Schaetzel SM, Price TP, Mandell KA, Ferrigno L, Salzberg M, DeUgarte DA, Kaji AH, Moran GJ, Saltzman D, Alam HB, Park PK, Kao LS, Thompson CM, Self WH, Yu JT, Wiebusch A, Winchell RJ, Clark S, Krishnadasan A, Fannon E, Lavallee DC, Comstock BA, Bizzell B, Heagerty PJ, Kessler LG, Talan DA. A Randomized Trial Comparing Antibiotics with Appendectomy for Appendicitis. N Engl J Med. 2020 Nov 12;383(20):1907-1919. doi: 10.1056/NEJMoa2014320. Epub 2020 Oct 5. PMID 33017106
- [Derived] Serrano E, Voldal EC, Machado-Aranda D, DeUgarte DA, Kao L, Drake T, Winchell R, Cuschieri J, Krishnadasan A, Talan DA, Siparsky N, Ayoung-Chee P, Self WH, McGonagill P, Mandell KA, Liang MK, Dodwad SJ, Thompson CM, Padilla RM, Fleischman R, Price TP, Jones A, Bernardi K, Garcia L, Evans HL, Sanchez SE, Odom S, Comstock BA, Heagerty PJ, Lawrence SO, Monsell SE, Fannon EEC, Kessler LG, Flum DR, Davidson GH; Writing Group for the CODA Collaborative. Trial Participation and Outcomes Among English-Speaking and Spanish-Speaking Patients With Appendicitis Randomized to Antibiotics: A Secondary Analysis of the CODA Randomized Clinical Trial. JAMA Surg. 2023 Sep 1;158(9):901-908. doi: 10.1001/jamasurg.2023.2277. PMID 37379001
- [Derived] Writing Group for the CODA Collaborative; Zhang IY, Voldal EC, Davidson GH, Liao JM, Thompson CM, Self WH, Kao LS, Cherry-Bukowiec J, Raghavendran K, Kaji AH, DeUgarte DA, Gonzalez E, Mandell KA, Ohe K, Siparsky N, Price TP, Evans DC, Victory J, Chiang W, Jones A, Kutcher ME, Ciomperlik H, Liang MK, Evans HL, Faine BA, Neufeld M, Sanchez SE, Krishnadasan A, Comstock BA, Heagerty PJ, Lawrence SO, Monsell SE, Fannon EEC, Kessler LG, Talan DA, Flum DR. Association of Patient Belief About Success of Antibiotics for Appendicitis and Outcomes: A Secondary Analysis of the CODA Randomized Clinical Trial. JAMA Surg. 2022 Dec 1;157(12):1080-1087. doi: 10.1001/jamasurg.2022.4765. PMID 36197656
- [Derived] Thompson CM, Voldal EC, Davidson GH, Sanchez SE, Ayoung-Chee P, Victory J, Guiden M, Bizzell B, Glaser J, Hults C, Price TP, Siparsky N, Ohe K, Mandell KA, DeUgarte DA, Kaji AH, Uribe L, Kao LS, Mueck KM, Farjah F, Self WH, Clark S, Drake FT, Fischkoff K, Minko E, Cuschieri J, Faine B, Skeete DA, Dhanani N, Liang MK, Krishnadasan A, Talan DA, Fannon E, Kessler LG, Comstock BA, Heagerty PJ, Monsell SE, Lawrence SO, Flum DR, Lavallee DC; Writing Group for the CODA Collaborative. Perception of Treatment Success and Impact on Function with Antibiotics or Appendectomy for Appendicitis: A Randomized Clinical Trial with an Observational Cohort. Ann Surg. 2023 Jun 1;277(6):886-893. doi: 10.1097/SLA.0000000000005458. Epub 2022 Jul 11. PMID 35815898
- [Derived] Writing Group for the CODA Collaborative; Talan DA, Moran GJ, Krishnadasan A, Monsell SE, Faine BA, Uribe L, Kaji AH, DeUgarte DA, Self WH, Shapiro NI, Cuschieri J, Glaser J, Park PK, Price TP, Siparsky N, Sanchez SE, Machado-Aranda DA, Victory J, Ayoung-Chee P, Chiang W, Corsa J, Evans HL, Ferrigno L, Garcia L, Hatch Q, Horton MD, Johnson J, Jones A, Kao LS, Kelly A, Kim D, Kutcher ME, Liang MK, Maghami N, McGrane K, Minko E, Mohr C, Neufeld M, Patton JH, Rog C, Rushing A, Sabbatini AK, Salzberg M, Thompson CM, Tichter A, Wisler J, Bizzell B, Fannon E, Lawrence SO, Voldal EC, Lavallee DC, Comstock BA, Heagerty PJ, Davidson GH, Flum DR, Kessler LG. Analysis of Outcomes Associated With Outpatient Management of Nonoperatively Treated Patients With Appendicitis. JAMA Netw Open. 2022 Jul 1;5(7):e2220039. doi: 10.1001/jamanetworkopen.2022.20039. PMID 35796152
- [Derived] Writing Group for the CODA Collaborative; Davidson GH, Monsell SE, Evans H, Voldal EC, Fannon E, Lawrence SO, Krishnadasan A, Talan DA, Bizzell B, Heagerty PJ, Comstock BA, Lavallee DC, Villegas C, Winchell R, Thompson CM, Self WH, Kao LS, Dodwad SJ, Sabbatini AK, Droullard D, Machado-Aranda D, Gibbons MM, Kaji AH, DeUgarte DA, Ferrigno L, Salzberg M, Mandell KA, Siparsky N, Price TP, Raman A, Corsa J, Wisler J, Ayoung-Chee P, Victory J, Jones A, Kutcher M, McGrane K, Holihan J, Liang MK, Cuschieri J, Johnson J, Fischkoff K, Drake FT, Sanchez SE, Odom SR, Kessler LG, Flum DR. Self-selection vs Randomized Assignment of Treatment for Appendicitis. JAMA Surg. 2022 Jul 1;157(7):598-608. doi: 10.1001/jamasurg.2022.1554. PMID 35612859
- [Derived] Davidson GH, Flum DR, Talan DA, Kessler LG, Lavallee DC, Bizzell BJ, Farjah F, Stewart SD, Krishnadasan A, Carney EE, Wolff EM, Comstock BA, Monsell SE, Heagerty PJ, Ehlers AP, DeUgarte DA, Kaji AH, Evans HL, Yu JT, Mandell KA, Doten IC, Clive KS, McGrane KM, Tudor BC, Foster CS, Saltzman DJ, Thirlby RC, Lange EO, Sabbatini AK, Moran GJ. Comparison of Outcomes of antibiotic Drugs and Appendectomy (CODA) trial: a protocol for the pragmatic randomised study of appendicitis treatment. BMJ Open. 2017 Nov 15;7(11):e016117. doi: 10.1136/bmjopen-2017-016117. PMID 29146633

RESULTS

PARTICIPANT FLOW:
Groups:
- Antibiotics Therapy Arm: Patients in the antibiotics (abx) arm will receive a total of 10 days of abx, with a minimum of 24 hours using an IV abx formulation (administered in q8, q12, or q24 hour regimens with or without concurrent oral abx) followed by oral abx for the remainder of the 10 days. Pts will be offered a treatment regimen of abx based on guidelines published jointly by the Surgical Infection Society and the Infectious Disease Society of America. Any of the IV abx options (Single antibiotic-Cefoxitin, Ertapenem, Moxifloxicin, Tigecycline, Ticarcillin-Clavulanic Acid or Dual antibiotics-Metronidazole plus one of the following-Cefazolin, Cefuroxime, Ceftriaxone, Cefotaxime, Ciprofloxacin, Levofloxacin) will be considered acceptable. After IV abx, a regimen of oral abx will be continued for a total treatment length of 10 days.
Period: Overall Study
Arm/Group | Antibiotics Therapy Arm | Appendectomy Arm
Started | 776 | 776
30 Day Follow up | 702 | 695
Completed | 676 | 656
Not Completed | 100 | 120

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Antibiotics Therapy Arm | Appendectomy Arm | Total
Number analyzed (Participants) | 776 | 776 | 1552
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 745 | 748 | 1493
  >=65 years | 31 | 28 | 59
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.3 (13.4) | 37.8 (13.7) | 38.1 (13.5)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender different from sex assigned at birth | 8 | 6 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 286 | 290 | 576
  Male | 490 | 486 | 976
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 13 | 9 | 22
  Asian | 39 | 53 | 92
  Native Hawaiian or Other Pacific Islander | 4 | 3 | 7
  Black or African American | 75 | 63 | 138
  White | 461 | 449 | 910
  More than one race | 176 | 185 | 361
  Unknown or Not Reported | 8 | 14 | 22
Region of Enrollment [Number; unit: participants]
  United States | 776 | 776 | 1552

OUTCOME MEASURES:

1. Primary Outcome: Patient-reported Quality of Life as Measured by EuroQol (EQ-5D)
Description: The primary evaluation of patient-reported quality of life, as measured by the EuroQuol-5D at four-weeks, will be conducted using an intention-to-treat (ITT) analysis, where patients' data are analyzed according to the patients' randomized treatment assignment. EQ5D assesses health status in terms of five dimensions of health. The maximum score of 1 indicates the best health state, the minimum score is 0 (as score as bad as being dead).
Time Frame: Four-weeks after randomization
Population: The overall number of participants in each arm represents the number of participants who responded to the EQ-5D questions on the 4 week survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Antibiotics Therapy Arm | Appendectomy Arm
Number analyzed (Participants) | 683 | 664
score on a scale | 0.92 (0.13) | 0.91 (0.13)

2. Secondary Outcome: Total Number of Patients Who Had Resolution of Appendicitis Symptoms at 30 Days
Description: Total Number of Patients who had resolution of appendicitis symptoms at 30 Days. This was measured as absence of fever and abdominal pain and tenderness.
Time Frame: at 30 days
Population: Patients in each arm are reflective of the total n (participants) who responded to the appendicitis symptoms questions in the 4 week survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Antibiotics Therapy Arm | Appendectomy Arm
Number analyzed (Participants) | 676 | 663
Participants | 462 | 466

3. Secondary Outcome: Rate of Participants With Perforated Appendicitis
Description: Rates of patients who had perforated appendicitis will be calculated for each arm among those received an appendectomy.
Time Frame: 90 days post enrollment
Population: Overall Number of Participants in each arm is reflective those participants who had surgery by 90 days post enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Antibiotics Therapy Arm | Appendectomy Arm
Number analyzed (Participants) | 185 | 621
Participants | 59 | 99

4. Secondary Outcome: Number of Participants With at Least One Complications From Treatment
Description: Comparison of the number of participants with at least one surgical complication and antibiotic complications.
Time Frame: 90 days
Population: Total n of participants in each arm is reflective of those participants who completed the 90 day survey.
Measure: Count of Participants; unit: Participants
Groups:
- Antibiotics Therapy Arm: Patients in the antibiotics (abx) arm will receive a total of 10 days of abx, with a minimum of 24 hours using an IV abx formulation (administered in q8, q12, or q24 hour regimens with or without concurrent oral abx) followed by oral abx for the remainder of the 10 days. Patients will be offered a treatment regimen of abx based on guidelines published jointly by the Surgical Infection Society and the Infectious Disease Society of America. Any of the IV abx options (Single antibiotic-Cefoxitin, Ertapenem, Moxifloxicin, Tigecycline, Ticarcillin-Clavulanic Acid or Dual antibiotics-Metronidazole plus one of the following-Cefazolin, Cefuroxime, Ceftriaxone, Cefotaxime, Ciprofloxacin, Levofloxacin) will be considered acceptable. After IV abx, a regimen of oral abx will be continued for a total treatment length of 10 days.
  C
Arm/Group | Antibiotics Therapy Arm | Appendectomy Arm
Number analyzed (Participants) | 676 | 656
Participants | 37 | 21

5. Secondary Outcome: Rates of Participants With Appendiceal Cancer
Description: Rates of appendiceal cancer among participants will be calculated among the antibiotics and appendectomy arms.
Time Frame: Through study completion, up to 2 years
Population: Total number of participants is reflective of participants randomized to each arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Antibiotics Therapy Arm | Appendectomy Arm
Number analyzed (Participants) | 776 | 776
Participants | 4 | 6

6. Secondary Outcome: Days in Hospital After Index Treatment Within 90 Days
Description: Mean number of days in the hospital per participant calculated at 90 days post randomization. (Number of days/Number of Participants in Therapy Arm who responded to the 90 day survey question)
Time Frame: 90 days post randomization
Population: Number of Participants in each arm is reflective of participants who completed the 90 day survey question regarding days in the hospital.
Measure: Mean (95% Confidence Interval); unit: Days per participant (rate)
Arm/Group | Antibiotics Therapy Arm | Appendectomy Arm
Number analyzed (Participants) | 622 | 609
Days per participant (rate) | 0.68 [-3.36 to 4.72] | 0.15 [-2.05 to 2.35]

7. Secondary Outcome: Number of Clinic Visits or Emergency Room Visits
Description: Total number of participants with any visit to emergency department or urgent care clinic after index treatment within 90 days
Time Frame: 90 days post randomization
Population: Number of Participants in each arm is reflective of participants who completed the 90 day survey question regarding clinic or emergency room visits.
Measure: Number; unit: visits
Arm/Group | Antibiotics Therapy Arm | Appendectomy Arm
Number analyzed (Participants) | 618 | 604
visits | 55 | 26

8. Secondary Outcome: Eventual Appendectomy Incidence Proportion
Description: incidence proportion of appendectomy within 90 days post randomization among those randomized to antibiotics
Time Frame: 90 days post randomization
Population: Total Number of participants randomized to antibiotics
Measure: Number (95% Confidence Interval); unit: incidence proportion
Arm/Group | Antibiotics Therapy Arm
Number analyzed (Participants) | 776
incidence proportion | 0.29 [0.26 to 0.32]

ADVERSE EVENTS:
Time Frame: Adverse events from enrollment to 90 days.
Description: Total number of participants at risk is reflective of number of participant who completed a survey at 90 days post randomization.
Arm/Group | Antibiotics Therapy Arm | Appendectomy Arm
All-Cause Mortality (participants affected / at risk) | 0/676 | 0/656
Serious Adverse Events (participants affected / at risk) | 19/676 | 19/656
Other Adverse Events (participants affected / at risk) | 26/676 | 5/656
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antibiotics Therapy Arm (N=676) | Appendectomy Arm (N=656)
Unplanned hospitalization not for appendectomy (General disorders) | 19 (27) | 19 (20)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antibiotics Therapy Arm (N=676) | Appendectomy Arm (N=656)
Reaction to antibiotics that led to a health care encounter (General disorders) | 22 (676) | 1 (656)
Clostridioides difficile colitis (General disorders) | 4 (4) | 4 (4) — Clostridioides difficile colitis

LIMITATIONS AND CAVEATS:
Almost all patients with appendicitis were approached,~30% of eligible patients agreed to undergo randomization, with variation across sites, and this factor may have introduced selection bias. As a pragmatic trial, the protocol did not specify requirements for hospitalization or for a given antibiotic regimen. The trial was not blinded. Some patients in the antibiotics group underwent appendectomy without meeting protocol-specified criteria for surgery

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT02800785/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT02800785/SAP_001.pdf